CLINICAL TRIAL: NCT07180823
Title: The LungVision Navigational Platform for Preoperative Labeling of Pulmonary Ground Glass Nodules With Fiducial Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Piero Candoli, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GGN_LungVision_Fiducial_Marker; RC-2024-2790060 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchoscopy with Lung Vision navigation system (Experimental): Augmented fluoroscopy will be used as a guidance tool, which is already in use at our operating unit as part of normal clinical practice, and will be combined with radial ultrasound using a mini probe. Once the peripheral lesion has been located, a cytological and histological sample will be taken using a needle and/or forceps and/or cryoprobe under augmented fluoroscopic guidance and with R-EBUS, as per normal current clinical practice. If atypical cells or malignant tumour cells are found during the extemporaneous cytological examination, the FM, acquired specifically for the study, will be positioned to mark the pulmonary nodule. A coil-tailed FM will be used. Enhanced fluoroscopy will be used via the LungVision system.
  Interventions: Device: Bronchoscopy with Lung Vision navigation system

INTERVENTIONS:
Device: Bronchoscopy with Lung Vision navigation system — The procedure begins with inspection of the airways up to the subsegmental branches using a flexible bronchoscope. During the procedure, augmented fluoroscopy will be used as a guidance tool, which is already in use at our operating unit as part of normal clinical practice, and will be combined with radial ultrasound using a mini probe. Once the peripheral lesion has been located, a cytological and histological sample will be taken using a needle and/or forceps and/or cryoprobe under augmented fluoroscopic guidance and with R-EBUS, as per normal current clinical practice. If atypical cells or malignant tumour cells are found during the extemporaneous cytological examination, the FM, acquired specifically for the study, will be positioned to mark the pulmonary nodule. A coil-tailed FM will be used. Enhanced fluoroscopy will be used via the LungVision system.

SUMMARY:
Based on current evidence, there are no studies investigating the possibility of placing a fiducial marker using augmented fluoroscopy, particularly for partially solid lesions that are often not visible on traditional fluoroscopy. The study in question could provide evidence that will allow, in the future, the use of the LungVision system and radial ultrasound to effectively mark a lesion with a ground glass component highly suspected of malignancy via bronchoscopy, avoiding more invasive marking procedures such as trans-thoracic marking. Correct marking of the target lesion will allow easy identification of the lesion during surgery and its complete removal through small resections, obtaining a definitive histological diagnosis and, in some cases, radical oncological treatment with preservation of healthy lung tissue.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related deaths, accounting for 1.8 million deaths in 2020. For this reason, early screening, diagnosis and treatment play a crucial role in improving the survival rate of lung cancer patients. The cyto-histological typing of peripheral lung nodules can be performed percutaneously (transcutaneous ultrasound or CT-guided biopsy) or bronchoscopically. The CT-guided transcutaneous biopsy approach has a diagnostic yield of over 90%, but carries a high risk of pneumothorax (up to ¼ of cases), which requires chest drainage in up to 5% of cases. The bronchoscopic approach reduces the risk of complications, but the diagnostic yield is significantly lower, ranging from 34% to 63%. The yield of the bronchoscopic approach depends on the size of the lesion (further reduced if less than 20 mm), the presence of an afferent bronchus to the nodule (bronchus sign), the location of the nodule and the experience of the operator. The LungVision system is a navigation system based on augmented fluoroscopy which, using artificial intelligence algorithms, improves the visualisation, localisation and sampling of lung nodules. The system integrates high-resolution computed tomography (HRCT) acquired pre-procedurally with real-time fluoroscopic scans during the procedure to assist the operator in locating and sampling the lesion. Overall, according to the data currently available in the literature, derived mainly from three clinical studies, a high percentage of lesion localisation (between 80 and 94.7%), a diagnostic yield varying between 75 and 87.7% and a high safety profile are reported. Attempts to biopsy the solid component of these nodules in the preoperative phase are often unfeasible or inconclusive in the clinical setting. Currently, if malignancy is highly suspected, surgical biopsy using various localisation methods is recommended. Among the possible localisation methods are the so-called "fiducial markers". These are radiopaque instruments, usually small metal bars or micro-coils, which can be placed inside or near the target lesion to facilitate its localisation during surgical resection or stereotactic radiotherapy. Fiducial markers can be placed percutaneously under CT guidance, endovascularly or, as demonstrated by recent studies, even bronchoscopically using various guidance methods safely and effectively. Bronchoscopic FM placement also offers certain advantages, including the possibility of performing biopsies on lung nodules or lymph nodes during the same session and managing any intra-procedural bleeding. Among the future prospects, one of the possible fields of application of bronchoscopic navigation associated with augmented fluoroscopy could be the placement of fiducial markers for ground glass lesions, which are often not visible with traditional fluoroscopy, given the possibility of verifying the three-dimensional location of the bronchoscope or guide catheter in relation to the target lesion (tool-in-lesion). This would avoid positioning via a more invasive route or one with a higher risk of complications, such as the transthoracic route. For these reasons, it has been hypothesised that the LungVision system, combined with radial endobronchial ultrasound, currently in use in the clinical practice of the Interventional Pulmonology Unit, could be used to locate peripheral lung lesions with a ground-glass component and place a cs-FM via bronchoscopy in the preoperative phase. This would confirm the possibility of placing the FM using the LungVision system combined with radial ultrasound, allowing for subsequent surgical removal and definitive histological typing of the target lesion.

Uncontrolled, monocentric interventional study, to be considered exploratory. Patients who meet the inclusion criteria and have given their informed consent will be enrolled consecutively. No blinding is planned. Patients will undergo bronchoscopy for cytohistological typing of GGN using a needle and/or forceps and/or cryoprobe under radial ultrasound and augmented fluoroscopic guidance, followed by immediate cytological examination in accordance with the normal clinical practice of the operating unit. In the event of cellular atypia or malignant tumour cells, the CT-FM will be placed under augmented fluoroscopic and radial ultrasound guidance to locate and mark the target lung lesion. If the immediate cytological examination is negative, the patient will be excluded from the study. If it is not possible to locate the target lesion using augmented fluoroscopy, the patient will be discharged from the study. On the same day, a chest CT scan will be performed to check the positioning of the FM. The day after the bronchoscopic procedure, the patient will undergo surgery to resect the lung lesion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Evidence of a partially solid peripheral pulmonary nodule with a solid component ≥ 6 mm or increasing in size, even if smaller, with a bronchus sign or adjacent bronchus on chest CT;
* Obtaining the patient's informed consent.

Exclusion Criteria:

* Pregnancy or suspected pregnancy;
* Contraindication to performing bronchoscopy under deep sedation, based on the anesthesiologist's assessment;
* Patient not eligible for surgery due to high surgical risk, based on the anesthesiologist's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visualisation (%) of the displacement catheter at the target lesion after 3D reconstruction by the LungVision system software | During the bronchoscopy procedure
  Investigate the possibility of reaching the target lung lesion with a fiducial marker displacement catheter, using the Lung Vision System's 'tool in lesion' feature as verification.
Percentage of lung lesions + fiducial markers removed out of the total number of lung lesions undergoing surgery | During the final post-surgical histological examination (up to 1 month post surgery)
  Describe the ability to completely resect the ground glass lung lesion marked with a fiducial marker
Number of lung lesions surgically resected with disease-free surgical margins out of the total number of lung lesions resected | During the final post-surgical histological examination (up to 1 month post surgery)
  Calculate the percentage of disease-free surgical resection margins out of all procedures performed.
Complication rate (overall and by type: pneumothorax, FM migration, hemoptysis) within one month of surgery. | During the endoscopic procedurePost-operatively (up to 1 month post surgery)At the telephone follow-up one month after surgery
  Calculate the frequency and type of complications related to fiducial marker placement.

SECONDARY OUTCOMES:
Time to navigate to the target nodule (minutes) Time to place the fiducial marker (minutes) | During the endoscopic procedure
  Describe the technical times required for navigation to the lesion and placement of the fiducial marker.
Distance between: -fiducial marker and target lesion -fiducial marker and resection margins -target lesion and resection margins -target lesion and pleura -fiducial marker and pleura | During histological examination of the surgical specimen (up to 1 month post surgery)
  Assess the effectiveness of fiducial marker placement also in relation to the position of the target lesion with respect to the pleura.
Time elapsed in the operating room between the start of the search for the fiducial marker using fluoroscopy and the end of the surgical resection | During the surgical procedure
  Describe the time required to locate the fiducial marker in the operating room.
Proportion of lesions in which the fiducial marker is visible with intraoperative ultrasound, calculated as: (n of fiducial markers visible with intraoperative ultrasound) / n total fiducial markers | During the surgical procedure
  Exploring the possibility of recognizing the fiducial marker with an intraoperative ultrasound scanner

CONTACTS AND LOCATIONS:
Overall Officials: Piero Candoli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy